CLINICAL TRIAL: NCT00757068
Title: Addressing Postpartum Mood and Weight Concerns to Sustain Smoking Cessation
Brief Title: Strategies to Avoid Returning to Smoking
Acronym: STARTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEVINER01; R01DA021608 (NIH)
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Smoking
Keywords: Non-smoking; Women; Pregnancy; Treatment; Mood; Weight; Supportive; Adjustment
MeSH Terms: conditions — Smoking; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SBT (Active Comparator): Women assigned to SBT (blue) will receive a six month program that offers to help them stay quit after having a baby.
  Interventions: Behavioral: Supportive Behavioral Therapy
- CBT (Experimental): Women assigned to CBT (pink) will receive a six month treatment designed to provide support and address the concerns of women who have just had a baby and do not want to resume smoking.
  Interventions: Behavioral: CBT addressing postpartum mood and weight concerns

INTERVENTIONS:
Behavioral: CBT addressing postpartum mood and weight concerns — Women will be assigned an individual counselor who will meet with them face-to-face six times and telephone them seven times. In these treatment sessions, the counselor will address postpartum mood and weight concerns.
  Other Names: STARTS; Strategies to Avoid Returning to Smoking
  Arms: CBT
Behavioral: Supportive Behavioral Therapy — Women will be assigned an individual counselor who will meet with them face-to-face six times and telephone them seven times. A non-specific, supportive condition will be delivered to women who want to remain smoke-free after they give birth.
  Other Names: Smoking cessation; General
  Arms: SBT

SUMMARY:
The purpose of this study is to evaluate the relative efficacy of a postpartum smoking relapse prevention program, Strategies to Avoid Returning to Smoking (STARTS), and a supportive, nondirective comparison condition (SUPPORT) to increase the proportion of women who remain abstinent through 12 months postpartum. We hypothesize that women randomized to STARTS will maintain higher rates of smoking abstinence at 6 and 12 months postpartum, and expect STARTS to increase the length of time abstinence is sustained relative to SUPPORT.

DETAILED DESCRIPTION:
The goal of the proposed investigation is to determine whether a cognitive behavioral relapse prevention intervention designed to address mood and weight concerns during the postpartum period will decrease the rate of postpartum relapse to smoking. We propose a two-group, randomized controlled trial. Women who quit smoking as a result of pregnancy, have been quit for at least one month prior to delivery and are motivated to remain abstinent postpartum will complete baseline assessments and be randomly assigned during the third trimester of pregnancy to either a cognitive behavioral relapse prevention intervention specifically designed for women who quit smoking during pregnancy, Strategies to Avoid Returning To Smoking (STARTS), or a nonspecific, supportive condition (SUPPORT). Both conditions will receive written information on the dangers of postpartum smoking and an equivalent number and amount of sessions immediately prior to delivery and during the first six months postpartum. Women will be treated for the first six months postpartum because substantial evidence has shown the risk of relapse to be greatest during the six months immediately following delivery (McBride et al., 1990; Mullen et al., 1990). All women will complete assessments at baseline (during pregnancy) and 3, 6 and 12 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Women will be eligible to participate if they:

  * report having smoked daily for at least one month during the 3 months prior to becoming pregnant;
  * smoked at least 10 cigarettes per day before quitting;
  * report no smoking in the four weeks prior to enrollment;
  * are not currently smoking as verified by a CO less than 8ppm;
  * are at least 'somewhat' motivated to remain abstinent postpartum and
  * are at least 14 years of age.

Exclusion Criteria:

* Women with current, acute psychiatric disorders, including other substance use problems and symptoms that warrant immediate treatment will be referred for care and excluded from this trial.
* Women with psychiatric disorders (e.g., depressive or anxiety disorders), who are not acutely suicidal and in whom the symptoms are not severe enough to preclude participation in a randomized trial, will be eligible to participate. However, women taking psychiatric medications that may affect the mediators of treatment, such as antidepressant, anxiolytic or weight control medications, will be excluded from participation.
* Women who endorse current suicidality will be discussed immediately with the consulting physician and referred to the psychiatric emergency room for further evaluation as indicated.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Abstinence at 12 months postpartum | through 12 months

SECONDARY OUTCOMES:
Explore factors associated with abstinence postpartum. | 0-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michele D Levine, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Levine MD, Emery RL, Kolko Conlon RP, Marcus MD, Germeroth LJ, Salk RH, Cheng Y. Depressive Symptoms Assessed Near the End of Pregnancy Predict Differential Response to Postpartum Smoking Relapse Prevention Intervention. Ann Behav Med. 2020 Jan 24;54(2):119-124. doi: 10.1093/abm/kaz026. PMID 31219152
- [Derived] Levine MD, Cheng Y, Marcus MD, Kalarchian MA, Emery RL. Preventing Postpartum Smoking Relapse: A Randomized Clinical Trial. JAMA Intern Med. 2016 Apr;176(4):443-52. doi: 10.1001/jamainternmed.2016.0248. PMID 26998789